CLINICAL TRIAL: NCT05503706
Title: Evaluation of the Antidandruff Effect of a Shampoo on Subjects With Dandruff and Slight Itching. Single-blind, Monocentric Study Realized Under Dermatological Control
Brief Title: Effects on the Scalp Lipids and TEWL of a 1% Selenium Disulfide and 1% Salicylic Acid Antidandruff Shampoo on Dandruff Scalp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ACR_VICO1BIS
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Dandruff
MeSH Terms: conditions — Dandruff | interventions — selenium disulfide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 1% Selenium Disulfide (SeS2)/1% salicylic acid-based shampoo — dandruff shampoo

SUMMARY:
The aim of this study was to investigate the changes in the scalp lipids and TEWL in dandruff subjects treated by 1% Selenium Disulfide (SeS2)/1% salicylic acid-based shampoo after an antidandruff treatment and after a remanence phase

DETAILED DESCRIPTION:
Dandruf often has a substantial negative impact on quality of life. The proliferation of Malassezia specie has been shown to be linked to dandruff. Yet, the sebum is essential for the growth of Malassezia restricta.

The sebum is mainly constituted by waxes, squalene and triglycerides. The triglycerides are partially transformed in free fatty acids while the squalene can be oxidized. Therefore, the change in lipids can be of interest for dandruff studies.

The scalp barrier function of a dandruff scalp is known to be altered and must recover after an antidandruff treatment

The aim of this study is to investigate the change of the scalp lipids and TEWL after a 1% selenium disulfide and 1% salicylic acid antidandruff shampoo on dandruff scalp and after a remanence period

ELIGIBILITY:
Inclusion Criteria:

* Subject with hair length > 2 cm.
* Subject exhibiting slight to severe dandruff state of scalp: Total dandruff score (adherent + non-adherent) ≥ 4 (ranging from 0 to 10) including and adherent dandruff score ≥ 2.5 (ranging from 0 to 5) and no limit for non-adherent dandruff score, after clinical examination 3 days after the last shampoo performed on D-3.
* Subject with slight itching state of scalp: score before shampoo ≥3 (ranging from 0 to 9,) 3 days after the last shampoo performed on D-3.
* Subject usually using a shampoo 3 times a week and accepting to follow this rate during the whole study period.
* Subject having stopped any possible antidandruff treatment at least 1 week prior to study pre-inclusion.
* Subject usually using anti-dandruff products.
* Subject agreeing not to use any other cosmetic product on the air (tonic,lacquer, gel, mousse) and not colouring or bleaching hair until the end of study

Exclusion Criteria:

* Main Inclusion Criteria:

  * Subject with hair length > 2 cm.
  * Subject exhibiting slight to severe dandruff state of scalp: Total dandruff score (adherent + non-adherent) ≥ 4 (ranging from 0 to 10) including and adherent dandruff score ≥ 2.5 (ranging from 0 to 5) and no limit for non-adherent dandruff score, after clinical examination 3 days after the last shampoo performed on D-3.
  * Subject with slight itching state of scalp: score before shampoo ≥3 (ranging from 0 to 9,) 3 days after the last shampoo performed on D-3.
  * Subject usually using a shampoo 3 times a week and accepting to follow this rate during the whole study period.
  * Subject having stopped any possible antidandruff treatment at least 1 week prior to study pre-inclusion.
  * Subject usually using anti-dandruff products.
  * Subject agreeing not to use any other cosmetic product on the air (tonic,lacquer, gel, mousse) and not colouring or bleaching hair until the end of study
* Main Non-Inclusion Criteria:

  * Subject who has skin marks on the scalp that could interfere with the assessment (pigmentation trouble, scar elements…).
  * Subject who has used topic treatment for the scalp (anti-dandruff, antihairloss) or corticosteroid treatment (per os or topical) during the last two weeks before the start of the study.
  * Subject who has used products for the scalp (dyeing, bleaching, permanent waving and straightening …) within the 2 weeks prior to the study.
  * Subject with personal history of allergy and/or particular reactivity to antidandruff products.
  * Subject with personal history of allergy and/or adverse reactions to cosmetic products containing surfactant agents (soaps, shower gel, conditioner …)
  * Subject who has taken a drug containing lithium, corticoids, during the last month; anti-histaminic, anti-fungal, non-steroidal anti-inflammatory or immunosuppressive drugs during the last 7 days.
  * Subject who has taken retinoid acid (local or per os) since less than 6 months.
  * Subject with cutaneous affection of the scalp (psoriasis, atopic dermatitis, seborrheic dermatitis, alopecia …).
  * Subject affected by serious, non-stabilized or progressive disease (according to the investigator) as diabetes, hypertension, hypothyroidism or hyperthyroidism which may influence the evolution of studied cutaneous state and morphology.
  * Subject affected by serious pathology (cancer, immune-depressed)
  * Subject who has undergone a surgical operation in the previous month of the study or having planned it during the study.
  * Subject, who has started, stopped or changed of hormonal treatment (including contraceptive pill) in the previous 6 weeks.
  * Pregnancy or breastfeeding during the last 6 months, ongoing or planned during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change of squame quantity during the antidandruff treatment | 1 month
  squame level clinical scoring evaluation (adherent squame, non-adherent squame and total squame).

SECONDARY OUTCOMES:
Evaluate the change in scalp barrier function and lipids (glycerides, free fatty acids, squalene and peroxidized squalene) after the antidandruff treatment | 1 month
  Trans epidermal barrier by instrumental evaluation and lipids by chromatography
Evaluation of the scalp barrier function | 1 month
  The evaluation of the scalp barrier function was done by Transepidermal Water Loss (TEWL) measurement.

CONTACTS AND LOCATIONS:
Overall Officials: AUDREY GUENICHE, PHD, Study Chair — L'Oreal
Locations (1):
- DERMSCAN, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: Undecided